CLINICAL TRIAL: NCT00551980
Title: Effectiveness of a Workplace Cognitive and Physical Program in Reducing Headache,Neck and Shoulder Pain in an Extensive Working Community. A Randomized Controlled Trial
Brief Title: The Efficacy of a Cognitive and Physical Intervention to Reduce Head and Muscle Pain in a Working Community
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Compagnia di San Paolo (Other); Turin, Italy (Other); Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other); Regione Piemonte (Other)
Responsible Party: Franco Mongini/ Professor and chairman, Unit of Headache and Facial Pain, Dept. of Clinical Pathophysiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1130SD2006.1911
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Migraine; Tension Type Headache; Cervical Pain
Keywords: Headache; Cervical Pain; Cognitive treatment; Relaxation; Exercise
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache; Neck Pain; Headache; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive and physical program (Experimental): Randomized group of workers of the same institution ( City of Turin, Italy).
  Interventions: Behavioral: Cognitive, Relaxation, Exercise Therapy
- Control group (No Intervention): Randomized group of workers of the same institution ( City of Turin, Italy).

INTERVENTIONS:
Behavioral: Cognitive, Relaxation, Exercise Therapy — The intervention consists of brief shoulder and neck exercises to be performed several times a day, a relaxation exercise and instructions of how to reduce hyperfunction of the craniofacial and cervical muscles during the day
  Arms: Cognitive and physical program

SUMMARY:
This study is a controlled, cluster randomised, interventional trial to evaluate the effectiveness of a workplace cognitive and physical program (Intervention), in reducing the frequency of head and neck pain in an extensive working population.

DETAILED DESCRIPTION:
Many studies were performed to assess the efficacy of non invasive physical interventions in the treatment of different types of headache and cervical pain. However the evidence on their effectiveness is still limited and the results of recent studies are conflicting.

In a previous non-randomized-controlled study in which the cognitive and physical programme was applied to a consistent number of office workers, a significant reduction of frequency of pain in the head and neck areas and of analgesic drug consumption was obtained. The present study was designed to confirm the data in a much more extensive working population and applying a randomised design.

The primary objective is to confirm the effectiveness of a workplace cognitive and physical programme (Intervention), in reducing the frequency of pain involving the head and neck area in a large working community using a randomized design.The Intervention consists of brief shoulder and neck exercises to be performed several times a day, a relaxation exercise and instructions of how to reduce parafunction and hyperfunction of the craniofacial and cervical muscles during the day.

Secondary objectives:

To confirm the effectiveness of the Intervention, in reducing the intensity of pain involving the head and neck area in a large working community using a randomized design.

To confirm the reduction in analgesic drugs consumption after the Intervention in a large working community using a randomized design.

To evaluate the persistence of the effectiveness of the Intervention after 12 months in a large working community using a randomized design.

Comparison(s): Group of employees that will receive a cognitive/physical programme (Intervention), compared to a similar group of employees that will not receive the Intervention (Controls); (frequency of headache and neck and shoulder pain).

ELIGIBILITY:
Inclusion Criteria:

* All the subjects employed at the Municipality of Turin at September, 2007 will be recruited.

Exclusion Criteria:

* Because of the pragmatic design, no exclusion criteria are required for this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2895 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Reduction in number of days per month with headache and shoulders pain after 6 months.Proportion of subjects with more than 4 days with headache and shoulder pain at the baseline that will have reduction in pain frequency of more than 50%, after 6 months | 6 months

SECONDARY OUTCOMES:
Headache index (Intensity x Frequency) after 6 and 12 months. Frequency of analgesic drug consumption after 6 and 12 months Frequency of headache and shoulder pain after 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Franco Mongini, Professor, Study Chair — University of Turin, Italy; Chantal Milani, DDS, Principal Investigator — University of Turin, Italy; Luca Ferrero, DDS, Principal Investigator — University of Turin, Italy; Alessandro Ugolini, DDS, Principal Investigator — University of Turin, Italy; Monica Sigaudo, DDS, Principal Investigator — University of Turin, Italy; Elisa Chiorino, Dr, Principal Investigator — University of Turin, Italy
Locations (1):
- Headache and Facial Pain Unit University of Turin, Torino, Italy

REFERENCES:
- [Derived] Mongini F, Evangelista A, Milani C, Ferrero L, Ciccone G, Ugolini A, Piedimonte A, Sigaudo M, Carlino E, Banzatti E, Galassi C. An educational and physical program to reduce headache, neck/shoulder pain in a working community: a cluster-randomized controlled trial. PLoS One. 2012;7(1):e29637. doi: 10.1371/journal.pone.0029637. Epub 2012 Jan 9. PMID 22253751